CLINICAL TRIAL: NCT04688801
Title: Ajuvant Chemotherapy and Immunotherapy in Patients With Esophageal, Esophageal- Gastric Junction Cancer With or Without Preoperative Chemotherapy With High Risk for Recurrence (N+ and/ or R1)
Brief Title: Ajuvant Chemotherapy and Immunotherapy in Patients With Esophageal, Esophageal- Gastric Junction Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ajuvant immunotherapy ZYP
Record Dates: First submitted 2020-11-15; First posted 2020-12-30 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Cancer; Gastroesophageal Cancer; Immunotherapy; Adjuvant
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Antineoplastic Agents; Immunotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy± Radiotherapy Group (Active Comparator): Chemotherapy± Radiotherapy is used as adjuvant therapy for high risk patients after surgery with or without neoadjuvant therapy.
  Interventions: Drug: Chemotherapy Drugs, Cancer
- Chemotherapy + Immunotherapy ± Radiotherapy Group (Experimental): Chemotherapy + Immunotherapy ± Radiotherapy is used as adjuvant therapy for high risk patients after surgery with or without neoadjuvant therapy.
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Chemotherapy Drugs, Cancer — Chemotherapy± Radiotherapy after surgery
  Arms: Chemotherapy± Radiotherapy Group
Drug: Immunotherapy — Chemotherapy + Immuonotherapy ± Radiotherapy after surgery
  Arms: Chemotherapy + Immunotherapy ± Radiotherapy Group

SUMMARY:
Surgery with or without neoadjuvant therapy is usually used as the treatment for resectable esophageal cancer or esophageal- gastric junction cancer. Patients who have a poor response to neoadjuvant therapy and have an incomplete (R1) resection or have metastatic lymph nodes in the resection specimen (N+) are especially at risk of recurrence, to continue with the chemotherapy± radiotherapy is often used in these cases. However, the overall survival is still poor. We designed a prospective randomized controlled tial to study whether immunotherapy could be used with chemotherapy after surgery to improve overall survival. The primary endpoint ofthe study is disease free survival, with secondary endpoints of overall survival, safety and toxicity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Histologically proven esophageal or EG-junction carcinoma (Siewert I-II). The heart and lung function can tolerate surgery. The cancer is resectable and incurable therapy will be perfomed.

Exclusion Criteria:

EG-junction carcinoma (Siewert III). M1 stage according to the current (8th) version of TNMclassification system. The heart and lung function can't tolerate surgery. R2 Resection Status.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival rate | 5 years after surgery
  disease free survival after surgery
overall survival rate | 5 years after surgery
  overall survival after surgery

SECONDARY OUTCOMES:
Rate of adverse events | within 6 months
  Rate of adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI- CTCAE v5.0)
Quality of Life （KPS or PS or QOL or EORTC QLQ C30） | 5 years after therapy
  Quality of Life （KPS or PS or QOL or EORTC QLQ C30）after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Shandong University, Jinan, Shandong, China